CLINICAL TRIAL: NCT03955679
Title: A Managed Access Program (MAP) Cohort Treatment Protocol to Provide AVXS-101 to Patients With a Genetic Diagnosis of Spinal Muscular Atrophy (SMA) With 1, 2 or 3 Copies of SMN2
Brief Title: AveXis Managed Access Program Cohort for Access to AVXS-101
Status: Approved for marketing | Type: Expanded Access
Sponsor: United BioSource, LLC (Industry)
Collaborators: AveXis, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AVXS-101-MAP-001
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; Gene replacement therapy; AVXS-101; Compassionate Use; Managed Access Program; MAP
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Zolgensma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Genetic: AVXS-101 — AVXS-101 is a non-replicating recombinant adeno-associated virus serotype 9 (AAV9) containing the human survival motor neuron (SMN) gene under the control of the cytomegalovirus (CMV) enhancer/chicken β-actin-hybrid promoter (CB). AVXS-101 will be administered as a one-time intravenous infusion over approximately 60 minutes. Dosage will be determined by the participants weight.

SUMMARY:
The purpose of this Cohort Treatment Protocol will allow access to AVXS-101 for eligible patients diagnosed with SMA.

DETAILED DESCRIPTION:
The purpose of this Cohort Treatment Protocol will allow access to AVXS-101 for eligible patients diagnosed with SMA.

The requesting Physician submits a request for access to drug (often referred to as Compassionate Use) to AveXis which is reviewed and approved by the medical team experienced with the drug and indication. The requesting Physician should refer to the latest Investigator's Brochure (IB) or approved label for overview of drug including: nonclinical and clinical experience, risk and benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SMA must satisfy both a. and b. of the following specified criteria:

   1. Diagnosis of SMA based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and 1, 2, or 3 copies of SMN2.
   2. Either patients with onset of symptoms prior to < 6 months (< 180 days) of age or pre-symptomatic patients, less than 6 months of age, with 1, 2, or 3 copies of SMN2 who are not excluded for other reasons.
2. Weight ≥ 2.6 kg to ≤ 13.5 kg at dosing.
3. Patients must have a pre-treatment swallowing evaluation test performed prior to administration of AVXS-101.
4. Patients must have a formal pulmonary evaluation including documentation of non-invasive ventilatory use prior to administration of AVXS-101. Ventilation should be actively managed by an appropriately trained specialist per the published standard of care.
5. Up-to-date on childhood vaccinations. Seasonal vaccinations and palivizumab prophylaxis (also known as Synagis) to prevent respiratory syncytial virus (RSV) infections have been administered as recommended by the American Academy of Pediatrics.
6. Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with study procedures and visit schedule.

Exclusion Criteria:

1. Tracheostomy.
2. Contraindication to receiving glucocorticosteroids or their excipients.
3. Anti Adeno Associated Virus Serotype 9 (AAV9) antibody titer > 1:50 (or any value reported as elevated for the laboratory) as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay. Should a potential patient demonstrate AntiAAV9 antibody titer > 1:50, he or she may be retested and will be eligible to participate if the AntiAAV9 antibody titer upon retesting is ≤ 1:50.
4. Clinically significant abnormal laboratory values for troponin-I, and platelets. ALT, AST, bilirubin or gamma glutamyl transferase (GGT) > 2 x the upper limit of normal (ULN) prior to gene replacement therapy that in the judgment of the Treating Physician or AveXis would create too great a risk for the patient to be treated with AVXS-101 or prophylactic prednisolone. Note: Elevated bilirubin > 2 x ULN if associated with neonatal jaundice is not considered exclusionary.
5. Medical conditions, diagnoses (especially cardiac), or on concurrent medications prior to gene replacement therapy that in the judgment of the treating physician or sponsor would create too great a risk for the patient to be treated with AVXS-101 or prophylactic prednisolone.
6. Participation or expected participation in current treatment clinical study (with the exception of observational cohort studies or non-interventional studies) for an unapproved investigational agent.
7. Parent(s)/legal guardian(s) unwilling to keep study results/observations confidential or to refrain from posting confidential study results/observations on social media sites.
8. Parent(s)/legal guardian(s) refuses to sign consent form.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Mercuri E, Finkel RS, Muntoni F, Wirth B, Montes J, Main M, Mazzone ES, Vitale M, Snyder B, Quijano-Roy S, Bertini E, Davis RH, Meyer OH, Simonds AK, Schroth MK, Graham RJ, Kirschner J, Iannaccone ST, Crawford TO, Woods S, Qian Y, Sejersen T; SMA Care Group. Diagnosis and management of spinal muscular atrophy: Part 1: Recommendations for diagnosis, rehabilitation, orthopedic and nutritional care. Neuromuscul Disord. 2018 Feb;28(2):103-115. doi: 10.1016/j.nmd.2017.11.005. Epub 2017 Nov 23. PMID 29290580
- [Background] Finkel RS, Mercuri E, Meyer OH, Simonds AK, Schroth MK, Graham RJ, Kirschner J, Iannaccone ST, Crawford TO, Woods S, Muntoni F, Wirth B, Montes J, Main M, Mazzone ES, Vitale M, Snyder B, Quijano-Roy S, Bertini E, Davis RH, Qian Y, Sejersen T; SMA Care group. Diagnosis and management of spinal muscular atrophy: Part 2: Pulmonary and acute care; medications, supplements and immunizations; other organ systems; and ethics. Neuromuscul Disord. 2018 Mar;28(3):197-207. doi: 10.1016/j.nmd.2017.11.004. Epub 2017 Nov 23. PMID 29305137
- [Background] Committee on Infectious Diseases. From the American Academy of Pediatrics: Policy statements--Modified recommendations for use of palivizumab for prevention of respiratory syncytial virus infections. Pediatrics. 2009 Dec;124(6):1694-701. doi: 10.1542/peds.2009-2345. Epub 2009 Sep 7. PMID 19736258
- [Background] Mendell JR, Al-Zaidy S, Shell R, Arnold WD, Rodino-Klapac LR, Prior TW, Lowes L, Alfano L, Berry K, Church K, Kissel JT, Nagendran S, L'Italien J, Sproule DM, Wells C, Cardenas JA, Heitzer MD, Kaspar A, Corcoran S, Braun L, Likhite S, Miranda C, Meyer K, Foust KD, Burghes AHM, Kaspar BK. Single-Dose Gene-Replacement Therapy for Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1713-1722. doi: 10.1056/NEJMoa1706198. PMID 29091557
- [Background] Fu H, Meadows AS, Pineda RJ, Kunkler KL, Truxal KV, McBride KL, Flanigan KM, McCarty DM. Differential Prevalence of Antibodies Against Adeno-Associated Virus in Healthy Children and Patients with Mucopolysaccharidosis III: Perspective for AAV-Mediated Gene Therapy. Hum Gene Ther Clin Dev. 2017 Dec;28(4):187-196. doi: 10.1089/humc.2017.109. Epub 2017 Oct 24. PMID 29064732
- See also: Kroger A, Duchin J, Vazquez M. General Best Practice Guidelines for Immunization (ACIP). Accessed on 2018. — http://www.cdc.gov/vaccines/hcp/acip-recs/general-recs/downloads/general-recs.pdf